CLINICAL TRIAL: NCT01580241
Title: Expression Patterns of Stem Cell Marker Doublecortin and CaM Kinase-Like-1 (DCAMKL-1) in Human Pancreatic Adenocarcinoma
Brief Title: Serum DCAMKL1 Pre and Post Treatment in Patients With Pancreatic Cancer
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Other Study IDs: 2606
Record Dates: First submitted 2012-04-17; First posted 2012-04-18 (Estimated); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Surgery group: Patients with pancreatic cancer who undergo surgical treatment only
- Chemotherapy group: Patients with pancreatic cancer who undergo chemotherapy treatment only
- Neoadjuvant group: Patients with pancreatic cancer who undergo neoadjuvant chemotherapy and surgery
- Adjuvant group: Patients with pancreatic cancer who undergo surgery followed by chemotherapy

SUMMARY:
The investigators believe DCAMKL-1 is a stem cell tumor marker and is elevated in patients with pancreatic cancer. The investigators would like to analyze its expression pre and post treatment, to gauge the correlation between current pancreatic cancer therapies and the expression of DCAMKL-1

DETAILED DESCRIPTION:
Pancreatic adenocarcinoma has the worst prognosis of any major malignancy with a 3% 5 year survival. Major obstacles in treating pancreatic cancer include extensive local invasion and early metastasis. The incidence of pancreatic adenocarcinoma (PAC) has been increasing steadily. Epithelial-mesenchymal transition (EMT) plays a key role in cancer invasion and metastasis. Recently, a direct link between EMT and the gain of epithelial stem cell properties has been described. We have recently determined that DCAMKL-1, a microtubule-associated kinase expressed in post mitotic neurons, is a putative intestinal stem cell marker. We have also demonstrated that DCAMKL-1, a protein expressed in both normal stem cells and in cancer, likely promotes tumorigenesis through the regulation of pri-let-7a microRNA and c-Myc. We have recently demonstrated evidence that DCAMKL-1 is a marker for pancreatic cancer stem cells in surgical specimens. This study will investigate expression of DCAMKL-1 in pancreatic tissue obtained through EUS-FNA. Furthermore expression of DCAMKL-1 will also be investigated in serum obtained simultaneously.

ELIGIBILITY:
Inclusion Criteria:

* pancreatic cancer

Exclusion Criteria:

* age < 18, history of other types of cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Human patients with pancreatic cancer undergo various treatments for pancreatic cancer. We will examine the expression of Dcamkl-1 pre and post therapy (including, chemotherapy only, surgery only, neoadjuvant and adjuvant therapies) to correlate treatment with a change in DCAMKl-1 expression.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2010-10 (Actual); Primary Completion 2015-07 (Actual); Study Completion 2024-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Courtney Houchen, MD, Principal Investigator — University of Oklahoma
Locations (1):
- Stephensen Cancer Center, Oklahoma City, Oklahoma, United States